CLINICAL TRIAL: NCT05076500
Title: Investigating the Tumour Immune Response of Radiotherapy
Acronym: TIMM-RAD
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tim Illidge, Professor of Targeted Therapy and Oncology, University of Manchester
Other Study IDs: NHS001688; 21-XTEAM-13 (Other: Christie NHS Foundation Trust)
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pre-treatment and during/post-treatment tumour tissue, and matched blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Cervical cancer: Cervical cancer patients receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection
- Rectal cancer: Rectal cancer patients receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection
- Head and neck cancer: Head and neck cancer patients receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection
- nodal non-Hodgkin lymphoma: Patients with nodal NHL receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection
- cutaneous lymphoma: Patients with cutaneous lymphoma receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection
- cutaneous squamous cell carcinoma and basal cell carcinoma: Patients with cSCC and cBCC receiving standard of care radiotherapy
  Interventions: Procedure: Biopsy and blood sample collection

INTERVENTIONS:
Procedure: Biopsy and blood sample collection — A pre-treatment diagnostic biopsy sample plus 1 mandatory biopsy (during/post-radiotherapy [irradiated site]) will be collected from each participant.
  Matched blood samples will be collected from participants at baseline, during/post-radiotherapy, and if radiotherapy continues after the on-treatment biopsy is taken, an additional end of treatment blood sample will be collected.

SUMMARY:
This study aims to investigate immune changes which occur before and following standard radiotherapy in a range of tumour types. We will collect tissue and blood samples before and after radiation treatment from participants across six cancer types: cervical, rectal, Head and Neck cancer, nodal non-Hodgkin lymphoma, cutaneous lymphoma and cutaneous squamous cell carcinoma/ basal cell carcinoma.

DETAILED DESCRIPTION:
The purpose of this prospective, non-CTIMP, translational study is to assess the feasibility of achieving paired biopsies for immune analysis in patients across six different cancer types: cervical, rectal, Head and Neck cancer, nodal non-Hodgkin lymphoma, cutaneous lymphoma and cutaneous squamous cell carcinoma/ basal cell carcinoma.

All participants will have a minimum of 1 mandatory biopsy (during/post-radiotherapy [irradiated site]) and the potential to have a pre-treatment biopsy if the archival biopsy does not meet the suitability criteria.

Matched blood samples will be collected from participants at baseline, during/post-radiotherapy, and if radiotherapy continues after the on-treatment biopsy is taken, an additional end of treatment blood sample will be collected.

We aim to recruit 10-20 participants per study arm, with the option to increase numbers in study arms that are recruiting well - a maximum of 120 patients in total will be recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer, Stage I-IV, in one of the following: Cervical, rectal, nodal Non-Hodgkin lymphoma, cutaneous lymphoma, Head & neck cancer
* Diagnostic/pre-treatment biopsy confirmed suitable for translational research *
* Performance status - ECOG 0-2 (Refer to appendix 1), ECOG 3 allowed for arm F (unrelated to underlying cancer) as this group of patients often have ECOG 3 due to age and comorbidities.
* Age ≥ 18; no upper age limit.
* Participant considered suitable for radiotherapy
* Before participant registration, written informed consent must be given according to GCP and national regulations.

  *Pre-treatment biopsy must be from the gross tumour volume within the planned radiation field and must also:
* Have been formalin fixed for >12h and <72h
* Have tumour tissue and morphology confirmed by H&E staining
* Contain sufficient tumour cells (approximately 100)

Exclusion Criteria:

* Participants deemed unsuitable for a biopsy (during or following radiotherapy) in the opinion of the treating oncologist.
* Participants who have received chemotherapy within 28 days of starting radiotherapy.
* Participants with intercurrent or past history of hepatitis B, C or human immunodeficiency virus infection if known. A negative test result for hepatitis B, C and HIV infection is required prior to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtaining paired biopsy samples | Within 6-7 weeks of starting radiotherapy
  To assess the feasibility of obtaining tumour samples pre-radiotherapy (diagnostic or fresh) and a second biopsy during or immediately after radiotherapy, or a surgical sample, from patients undergoing standard of care RT.
Collection of matched blood samples | Within 6-7 weeks of starting radiotherapy
  To obtain additional matched blood samples pre-radiotherapy, during or post-radiotherapy, and at the end of radiotherapy for assessment of immune status of peripheral blood in comparison to the intratumoural microenvironment.

OTHER OUTCOMES:
Immunohistochemistry analysis of expression markers on tumour tissue | Within 6-7 weeks of starting radiotherapy
  Immunohistochemistry (IHC) analysis of expression markers on tumours pre-radiotherapy and during/post radiotherapy
RNA evaluation of immune signatures | Within 6-7 weeks of starting radiotherapy
  RNA evaluation of immune signatures in tumour tissue and blood pre-radiotherapy and during/post radiotherapy
Analysis of peripheral blood mononuclear cells | Within 6-7 weeks of starting radiotherapy
  Assessment of changes in immune phenotypic markers
Analysis of plasma proteins, cytokines and chemokines | Within 6-7 weeks of starting radiotherapy
  Analysis of plasma proteins, cytokines and chemokines as biomarkers of immune response

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Illidge, Study Chair — University of Manchester
Locations (1):
- Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No